CLINICAL TRIAL: NCT00941382
Title: Double-blind, Randomized Clinical Trial to Evaluate Effect of Combination Therapy of Metformin and Sibutramine Versus Metformin or Sibutramine Monotherapy Over Weight, Adiposity, Glucose Metabolism and Inflammatory State in Obese Patients
Brief Title: Sibutramine-metformin Combination Versus Sibutramine and Metformin Monotherapy in Obese Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Laboratorios Silanes S.A. de C.V. (Industry)
Responsible Party: Jorge González Canudas, Laboratorios Silanes S.A. de C.V.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OB Sil-02
Record Dates: First submitted 2009-07-14; First posted 2009-07-17 (Estimated); Last update posted 2009-07-17 (Estimated); Status verified 2009-07

CONDITIONS: Obesity
Keywords: sibutramine; metformin; obesity
MeSH Terms: conditions — Obesity | interventions — Combined Modality Therapy; sibutramine; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Sibutramin-Metformin (Experimental): Sibutramine-metformin therapy in a single tablet
  Interventions: Drug: Sibutramine-Metformin
- Sibutramine (Active Comparator): Sibutramine monotherapy
  Interventions: Drug: Sibutramine
- Metformin (Active Comparator): Metformin monotherapy
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Sibutramine-Metformin — sibutramine and metformin, 15 mg per day and 850 mg per day, respectively, in a single tablet, for 180 days
  Other Names: combination therapy
  Arms: Sibutramin-Metformin
Drug: Sibutramine — 15 mg per day for 180 days
  Other Names: Sibutramine monohidrate Hydrochloride
  Arms: Sibutramine
Drug: Metformin — Metformin 850 mg per day for 180 days
  Other Names: Metformin Hydrochloride
  Arms: Metformin

SUMMARY:
The aim of this study is to evaluate the effect of sibutramine and metformin combination therapy in comparison with sibutramine or metformin monotherapy over weight, adiposity, glucose metabolism and inflammatory state in obese patients.

DETAILED DESCRIPTION:
The treatment of obesity is strongly recommended because it exacerbates insulin resistance, hypertension, dyslipidemia and atherosclerosis, and represents a risk factor for type 2 diabetes. Although diet and exercise are valuable in this treatment, patient compliance is a major problem. Sibutramine has been shown to be a highly effective pharmacotherapy for weigh loss in obese patients, mediated by increased satiety and an enhancement of energy expenditure. Metformin is widely used for glycemia control and is associated with a small to moderate body weight loss. We are assessing the combination of sibutramine and metformin, two agents with different mechanisms of action for control of body weight and metabolic dysregulation.

ELIGIBILITY:
Inclusion criteria

* Age between 30 and 50 years
* Both genders
* BMI between 30 and 40
* Stable body weigh defined by over 5 per cent variability during the previous 3 months
* Fasting serum glucose less than 126 mg per dl
* Blood pressure over 140 and 90 mmHg
* Women ensuring contraceptive precautions.
* Communication and understanding capability.
* Informed consent awarding.

Exclusion criteria

* Women were excluded if they were pregnant or lactating potential while no taking adequate contraceptive precautions
* Any smoking during the preceding 6 months
* No physical activity, defined by less than 15 minutes per day of walking
* Excessive physical activity equivalent to running over 60 minutes per day
* Known hypersensitivity to sibutramine or metformin
* Low commitment to follow the protocol statements
* Any investigational medication during the preceding 6 months
* Any drug or substance mayor toxicity exposure during the preceding 3 months
* Alcohol or any drug abuse during the previous 3 months
* Current medication of oral corticosteroids, anticoagulants, sympathomimetics, sympatholytics, lipid lowering drugs, any medication for type 2 diabetes, and any sibutramine interaction drug
* Current or previous evidence of ischemic heart disease, cardiac arrhythmia, cerebrovascular disease, chronic hepatic disease, two fold persistent elevation of ALT, AST or FA
* Carrying a pacemaker or any permanent bioelectronic component that could interfere with bioimpedance process
* Renal failure defined by serum creatinine equal or ever 1.2 mg per dL
* Not controlled thyroid disease defined by altered serum T3, T4 and TSH during the previous 3 months
* Hypertension
* Type 2 diabetes
* Anti-depressants, or any psychiatric disturbance treatment

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-11; Primary Completion 2009-08 (Estimated); Study Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
improvement of body weight, adiposity and inflammation state defined by serum adiponectin, leptin and C reactive protein | 6 months

SECONDARY OUTCOMES:
improvement of metabolic profile, defined by triglycerides, total cholesterol, HDL cholesterol, LDL cholesterol, insulin, and insulin sensitivity | 6 months
adverse events | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jorge A González-Canudas, MD, Study Director — Laboratorios Silanes; Manuel González-Ortiz, PHD, Study Chair — University of Guadalajara; ESperanza Martínez-Abundis, PHD, Principal Investigator — University of Guadalajara
Locations (1):
- Centro Universitario de Ciencias de la Salud, Guadalajara, Jalisco, Mexico

REFERENCES:
- [Background] Cachofeiro V. Obesidad, Inflamación y disfunción endotelial. Rev Esp Obes 4: 194-204, 2006.
- [Background] Ferrannini E, Mari A. How to measure insulin sensitivity. J Hypertens. 1998 Jul;16(7):895-906. doi: 10.1097/00004872-199816070-00001. PMID 9794728
- [Background] Lyle WG; Plastic Surgery Educational Foundation DATA Committee. Pharmacological treatment of obesity. Plast Reconstr Surg. 2002 Nov;110(6):1577-80. doi: 10.1097/01.PRS.0000028331.84171.86. No abstract available. PMID 12409783
- [Background] Luque CA, Rey JA. The discovery and status of sibutramine as an anti-obesity drug. Eur J Pharmacol. 2002 Apr 12;440(2-3):119-28. doi: 10.1016/s0014-2999(02)01423-1. PMID 12007530
- [Background] Weigle DS. Pharmacological therapy of obesity: past, present, and future. J Clin Endocrinol Metab. 2003 Jun;88(6):2462-9. doi: 10.1210/jc.2003-030151. No abstract available. PMID 12788841
- [Background] Hundal RS, Inzucchi SE. Metformin: new understandings, new uses. Drugs. 2003;63(18):1879-94. doi: 10.2165/00003495-200363180-00001. PMID 12930161
- [Background] Bloomgarden ZT. Metformin. Diabetes Care. 1995 Jul;18(7):1078-80. doi: 10.2337/diacare.18.7.1078. No abstract available. PMID 7555549
- [Background] Campbell I. The obesity epidemic: can we turn the tide? Heart. 2003 May;89 Suppl 2(Suppl 2):ii22-4; discussion ii35-7. doi: 10.1136/heart.89.suppl_2.ii22. PMID 12695431
- [Background] McNulty SJ, Ur E, Williams G; Multicenter Sibutramine Study Group. A randomized trial of sibutramine in the management of obese type 2 diabetic patients treated with metformin. Diabetes Care. 2003 Jan;26(1):125-31. doi: 10.2337/diacare.26.1.125. PMID 12502668
- [Background] Love-Osborne K, Sheeder J, Zeitler P. Addition of metformin to a lifestyle modification program in adolescents with insulin resistance. J Pediatr. 2008 Jun;152(6):817-22. doi: 10.1016/j.jpeds.2008.01.018. Epub 2008 Mar 19. PMID 18492523
- [Background] Gonzalez-Ortiz M, Martinez-Abundis E, Mora-Martinez JM, Grover-Paez F. Renal handling of uric acid assessed by means of pharmacological tests in obese women. Diabetes Nutr Metab. 2001 Aug;14(4):189-94. PMID 11716287
- [Background] Clement K, Ferre P. Genetics and the pathophysiology of obesity. Pediatr Res. 2003 May;53(5):721-5. doi: 10.1203/01.PDR.0000059753.61905.58. Epub 2003 Mar 5. PMID 12621112
- [Background] Flegal KM, Carroll MD, Ogden CL, Johnson CL. Prevalence and trends in obesity among US adults, 1999-2000. JAMA. 2002 Oct 9;288(14):1723-7. doi: 10.1001/jama.288.14.1723. PMID 12365955
- [Background] Lozano Castañeda O. Adipocitoquinas. Rev Endocr Nutr. 10: 147-50, 2002.
- [Background] Karnehed N, Rasmussen F, Hemmingsson T, Tynelius P. Obesity and attained education: cohort study of more than 700,000 Swedish men. Obesity (Silver Spring). 2006 Aug;14(8):1421-8. doi: 10.1038/oby.2006.161. PMID 16988085
- [Background] Hensrud DD, Klein S. Extreme obesity: a new medical crisis in the United States. Mayo Clin Proc. 2006 Oct;81(10 Suppl):S5-10. doi: 10.1016/s0025-6196(11)61175-0. PMID 17036573